CLINICAL TRIAL: NCT03317119
Title: A Phase I Clinical Trial of Trametinib in Combination With TAS-102 in Patients With Chemotherapy-Resistant RAS-Mutated (PIK3CA/PTEN-Wild-Type) Metastatic Colorectal Cancer
Brief Title: Trametinib and Trifluridine and Tipiracil Hydrochloride in Treating Patients With Colon or Rectal Cancer That is Advanced, Metastatic, or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17212; NCI-2017-01923 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17212 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Colon Carcinoma; Metastatic Colorectal Carcinoma; Metastatic Rectal Carcinoma; RAS Family Gene Mutation; Stage III Colon Cancer AJCC v7; Stage III Colorectal Cancer AJCC v7; Stage III Rectal Cancer AJCC v7; Stage IIIA Colon Cancer AJCC v7; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIA Rectal Cancer AJCC v7; Stage IIIB Colon Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIB Rectal Cancer AJCC v7; Stage IIIC Colon Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IIIC Rectal Cancer AJCC v7; Stage IV Colon Cancer AJCC v7; Stage IV Colorectal Cancer AJCC v7; Stage IV Rectal Cancer AJCC v7; Stage IVA Colon Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVA Rectal Cancer AJCC v7; Stage IVB Colon Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7; Stage IVB Rectal Cancer AJCC v7
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — trametinib; Trifluridine; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TAS-102, trametinib) (Experimental): Patients receive trifluridine and tipiracil hydrochloride PO BID on days 1-5 and 8-12 and trametinib PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Trametinib; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: Lonsurf; TAS 102; TAS-102; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102

SUMMARY:
This phase I trial studies the side effects and best dose of trametinib and trifluridine and tipiracil hydrochloride in treating patients with colon or rectal cancer that has spread to other places in the body (advanced/metastatic) or cannot be removed by surgery. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as trifluridine and tipiracil hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving trametinib and trifluridine and tipiracil hydrochloride may prevent cancer cells from dividing and work better in treating patients with colon and rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) for the combination of trametinib and trifluridine and tipiracil hydrochloride (TAS-102) in patients with chemotherapy-resistant metastatic colorectal cancer.

SECONDARY OBJECTIVES:

I. Describe the safety of the combination of trametinib and TAS-102 across all investigated dose levels.

II. Describe the clinical activity including objective response rate (ORR), progression-free survival (PFS), and overall survival (OS) of the combination in an expansion cohort using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

OUTLINE:

Patients receive trifluridine and tipiracil hydrochloride orally (PO) twice daily (BID) on days 1-5 and 8-12 and trametinib PO once daily (QD) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then bi-annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* All patients must be able to take oral medications
* All patients must be deemed by investigator to have the initiative and means to be compliant with the study protocol (treatment and follow-up)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Pathologically confirmed advanced, unresectable, or metastatic colon or rectal cancer who have had intolerance to or progression after a fluoropyrimidine, oxaliplatin, irinotecan, and cetuximab or panitumumab in the event of wild-type RAS/BRAF tumors

  * Of note, prior bevacizumab or regorafenib exposure is not mandated as some patients are deemed poor candidates for anti-angiogenesis therapy and never receive these agents
* Tumors must have undergone expanded molecular profiling with a Clinical Laboratory Improvement Act (CLIA)-certified platform that evaluates, at a minimum, RAS, PIK3CA, PTEN and BRAF mutations status
* Documented RAS-mutated tumor without activating PIK3CA mutations or PTEN mutation (loss of PTEN or silencing)
* Measurable disease by RECIST 1.1 guidelines
* Last chemotherapy at least 3 weeks from initiation of study treatment
* No investigational agents within 4 weeks from initiation of study treatment
* Negative serum or urine beta-human chorionic gonadotropin (HcG) test (female patient of childbearing potential only) performed within 72 hours of prior to first study dose
* Absolute neutrophil count (ANC) >= 1500/mm^3 (to be performed within 28 days prior to day 1 of protocol therapy)

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 75,000/mm^3 without transfusions (to be performed within 28 days prior to day 1 of protocol therapy)
* Hemoglobin (Hgb) >= 8 g/dL without transfusions (to be performed within 28 days prior to day 1 of protocol therapy)
* Total serum bilirubin < upper limit of normal (ULN) (to be performed within 28 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 2.5 x ULN if no liver metastases or =< 5 x ULN if liver metastases (to be performed within 28 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 2.5 x ULN if no liver metastases or =< 5 x ULN if liver metastases (to be performed within 28 days prior to day 1 of protocol therapy)
* Creatinine < 1.5 x ULN or creatinine clearance of >= 60 mL/min per the Cockcroft-Gault formula (to be performed within 28 days prior to day 1 of protocol therapy)
* Female of childbearing potential: negative urine or serum pregnancy test (to be performed within 28 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Corrected QT (QTc) interval =< 480 ms (12 lead-electrocardiography [ECG]) (to be performed within 28 days prior to day 1 of protocol therapy)
* Left ventricular ejection fraction >= 50% as determined by multigated acquisition (MUGA) scan or echocardiogram (to be performed within 28 days prior to day 1 of protocol therapy)
* Normal eye examination (to be performed within 28 days prior to day 1 of protocol therapy)
* Women of childbearing potential must use highly effective methods of contraception throughout the study and for 4 months after study drug discontinuation
* Sexually active men must use a condom during intercourse while taking study drug and for 60 days after study drug discontinuation; a condom is required for vasectomized men to prevent delivery of study drug via seminal fluid

Exclusion Criteria:

* Prior chemotherapy, biologic, targeted, or radiotherapy within 3 weeks prior to entering study or not recovered from grade >= 2 adverse events (AEs) due to agents administered more than 4 weeks earlier (except alopecia or neuropathy)
* Prior MEK inhibitor or prior TAS-102 therapy
* Use of other investigational drugs
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity, or hypercoagulability syndromes)
* History of retinal degenerative disease
* History of Gilbert's syndrome
* Previous or concurrent malignancy with the following exceptions:

  * Adequately treated basal cell or squamous cell carcinoma of skin with adequate wound healing prior to study entry
  * In situ carcinoma of the cervix treated curatively and without evidence of recurrence
  * Primary malignancy completely resected and in complete remission >= 1 year
* History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass graft, coronary angioplasty, or stenting) < 6 months prior to screening
* Impaired cardiovascular function or clinically significant cardiovascular disease including any of the following: symptomatic congestive heart failure, clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening except for atrial fibrillation and paroxysmal supraventricular tachycardia
* Uncontrolled arterial hypertension despite appropriate medical therapy (systolic blood pressure > 160 or diastolic blood pressure > 100)
* Neuromuscular disorders associated with elevated creatine kinase (CK, e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, or spinal muscular atrophy)
* Started or planning to start on strenuous exercise regimen after first dose of study treatment (i.e., muscular activities, such as strenuous exercise, that can result in significant increase in plasma CK levels should be avoided while on trametinib treatment)
* Gastrointestinal (GI) disease or impairment of GI function (e.g., active ulcerative disease, uncontrolled nausea, vomiting, or diarrhea, malabsorption syndrome, or small bowel resection)
* Prior major surgery =< 3 weeks before study drug or not recovered from side effects of such procedure
* Ongoing grade >= 3 neuropathy
* Known hypersensitivity to any components of study drugs
* Prior intolerance to a fluoropyrimidine
* Any other condition that would, in the investigator's judgement, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medications, social/psychological issues, etc.)
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose defined for the combination of trametinib, and Trifluridine and Tipiracil Hydrochloride (TAS?102) as the highest dose level at which 0-1 out of 6 patients experience dose limiting toxicities | Up to 28 days
  Toxicities observed at each dose level will be categorized by type (organ affected or laboratory determination such as absolute neutrophil count), severity (by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] 4.0 and nadir or maximum values for the laboratory measures), time of onset (i.e., course number), duration, and reversibility or outcome.

SECONDARY OUTCOMES:
Incidence of adverse events assessed using NCI) CTCAE 4.0 | Up to 30 after last dose
  Will be summarized in terms of type and severity, along with dose modification/delays that resulted. Analysis will be primarily descriptive.
Objective response rate using Response Evaluation Criteria in Solid Tumor (RECIST) guideline, version 1.1 | Up to 1 year
Time to progression using RECIST guideline, version 1.1 | From start of treatment to time of progression or death, whichever occurs first, assessed up to 1 year
Overall survival | From start of treatment to death (any cause), assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marwan G Fakih, Principal Investigator — City of Hope Medical Center
Locations (8):
- United States (8):
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Mission Hills, Mission Hills, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope - Santa Clarita, Santa Clarita, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California

REFERENCES:
- [Derived] Chuang J, Gong J, Li SM, Wang C, Fakih M. A Phase I Clinical Trial of Trametinib in Combination with TAS-102 in Patients with Chemotherapy-Resistant RAS-Mutated (PIK3CA/PTEN-Wild Type) Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2022 Sep;21(3):252-258. doi: 10.1016/j.clcc.2022.05.004. Epub 2022 May 23. PMID 35738999